CLINICAL TRIAL: NCT03695224
Title: Association of Glaucoma Morbidity and Impairment of Topological Perception: a Cohort Study
Brief Title: Matching Glaucoma With Impaired Cognition
Acronym: MAGIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Xiulan Zhang, Director of Clinical Research Center, Sun Yat-sen University
Other Study IDs: 2018KYPJ126
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Morbidity of Primary Open Angle Glaucoma
Keywords: Topological perception; Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10 ml of whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Subjects with normal topological perception
  Interventions: Diagnostic Test: Topological perception test
- Group B: Subjects with abnormal topological perception
  Interventions: Diagnostic Test: Topological perception test

INTERVENTIONS:
Diagnostic Test: Topological perception test — Participants' topological perception are tested with self-designed devices. Participants are asked to respond to the figures shown on the screen, and a final score will appear after they finish all the questions.

SUMMARY:
Glaucoma is the leading cause of irreversible blindness in the world. The current study is designed to find the underlying relationship between impairment of topological perception and incidence of glaucoma.

DETAILED DESCRIPTION:
Glaucoma is currently the leading cause of irreversible blindness in the world. It has been a difficult task for ophthalmologists and researchers to diagnose glaucoma, especially in early stage. At present, glaucoma diagnosis mainly relies on OCT and visual field test, which have relatively low sensitivity and specificity at the early stage of glaucoma. Previous studies mainly focused on ocular manifestation of glaucoma. However, there was evidence that abnormalities of visual pathway also existed in patients with glaucoma, indicating cerebral cognitive defects may also be involved in glaucoma development. Thus, the current study was designed, in which subjects at high-risk of developing glaucoma are separated into two group based on test results of topological perception. After five years' follow-up, morbidity of primary open-angle glaucoma would be compared between groups to see if there was any relationship between impaired cognitive function and incidence of glaucoma.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18-55;
2. Best corrected visual acuity ≥ 0.6, capable of completing routine glaucoma examinations;
3. Spherical equivalent < 3D；
4. No history of other ocular diseases (except mild cataract), including diabetic retinopathy, age-related macular degeneration, optical neuropathy, eye trauma, strabismus, nystagmus, severe dry eye, ptosis of the eyelid, etc.

Exclusion Criteria:

1. Unable or unwilling to sign informed consent, or cannot comply with the study protocol
2. Diagnosed with any kind of glaucoma (based on visual field and OCT, etc) or primary angle-closure diseases(primary angle closure suspect and primary angle closure, based on gonioscopy and UBM examination);
3. History of ocular surgeries or laser;
4. Diagnosed with specific neurologic diseases or psychiatric disorders: Parkinson's disease, Alzheimer's disease, anxiety, depression, schizophrenia, etc.(based on scale screening)
5. With severe systemic diseases: diabetes mellitus, hypertension(systolic pressure≥160mmHg or diastolic pressure≥100mmHg ), heart diseases, kidney diseases, rheumatological disorder, digestive diseases, cancer, etc.
6. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from communities in Guangzhou and nearby cities. Subjects fulfilling the above eligibility criteria will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-10-08 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Morbidity of primary open-angle glaucoma | From October 2018 to September 2024
  Incidence of primary open angle glaucoma in the study subjects

SECONDARY OUTCOMES:
Change in biometric parameters of optic nerve and macular region | From October 2018 to September 2024
  Biometric parameters of optic nerve include retinal nerve fiber layer (RNFL) thickness, ganglion cell layer (GCL) thickness, ganglion cell complex (GCC) thickness, etc.
Change in visual field | From October 2018 to September 2024
  Mean Deviation (MD value)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No